CLINICAL TRIAL: NCT04698304
Title: Physician-initiated, Prospective, Multi-center，Observational Study: The Efficacy of Endovascular Treatment in Femoropopliteal Occlusive Disease (FPOD) With TransAtlantic InterSociety Consensus (TASC) C and D Lesions
Brief Title: The Efficacy of Endovascular Treatment in FPOD With TASC C and D Lesions
Status: Active, not recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Second Affiliated Hospital of Suzhou University (Other); Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology (Other); Chengdu University of Traditional Chinese Medicine (Other); First Affiliated Hospital of Zhejiang University (Other); Xiamen Cardiovascular Hospital, Xiamen University (Other); Shanghai Zhongshan Hospital (Other); Huashan Hospital (Other); Qingdao Haici Hospital (Other); First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Other Study IDs: The Oriental Study
Record Dates: First submitted 2020-12-19; First posted 2021-01-06 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Femoropopliteal Occlusive Disease
Keywords: Femoropopliteal Occlusive Disease; endovascular treatment; patency rate

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group A：TASC C lesion group: Multiple stenoses or occlusions totaling >15cm or recurrent stenoses or occlusions that need treatment after endovascular interventions (300 cases)
  Interventions: Procedure: endovascular treatment
- Group B：TASC D lesion with common femoral artery involved: Chronic total occlusions >20cm with common femoral artery involved (100 cases)
  Interventions: Procedure: endovascular treatment
- Group C：TASC D lesion with proximal popliteal artery involved: Chronic total occlusions >20cm with proximal popliteal artery involved (300 cases)
  Interventions: Procedure: endovascular treatment
- Group D：TASC D lesion with distal popliteal artery involved: Chronic total occlusions >20cm with distal popliteal artery involved (200 cases)
  Interventions: Procedure: endovascular treatment
- Group E：TASC D lesion with popliteal artery and proximal trifurcation vessels involved: Chronic total occlusion of popliteal artery (P1-3 segment) with proximal trifurcation vessels involved (100 cases)
  Interventions: Procedure: endovascular treatment

INTERVENTIONS:
Procedure: endovascular treatment — All the patients are treated by endovascular therapy, through contralateral femoral artery approach, ipsilateral antegrade femoral artery approach or brachial artery approach. If the lesion is difficult to pass in antegrade approach, retrograde puncture at the distal artery of the lesion can be performed. Surgeons can choose treatment methods according to the characteristics of the lesions. For example: (a) Plain old balloon angioplasty; (b) Drug-coated balloon angioplasty; (c) Drug-coated balloon angioplasty + provisional stenting; (d) Bare-metal stent implantation; (e) Stent graft implantation; (f) Directional atherectomy + drug-coated balloon angioplasty, (g) Drug -eluting stent.

SUMMARY:
Based on the development of new tools, including drug coated balloon, paclitaxel eluting stent, interwoven stents, debulking tools, more challenging femoropopliteal arterial lesions have been treated with endovascular procedures.

The TASC D lesion ,especially with popliteal artery involved are often excluded in prospective clinical trials. Therefore, a well-designed real world study that track clinical relevant outcomes, are required to determine the optimal therapies for patients with complex femoropopliteal lesions.

DETAILED DESCRIPTION:
According to the TASC II guidelines, TASC D lesions was recommended for primary endovascular revascularization, TASC C lesions for surgical revascularization in patients with appropriate perioperative risk and available conduit. However, Based on the development of new tools, including drug coated balloon, paclitaxel eluting stent, interwoven stents, debulking tools, more challenging femoropopliteal arterial lesions have been treated with endovascular procedures.

Despite The shift of Endovascular- first strategy has been documented in recent literature. There still lack evidence to support either approach have a significant advantage over the other. And TASC D lesion ,especially with popliteal artery involved are often excluded in prospective clinical trials. Therefore, a well-designed real world study that track clinical relevant outcomes, are required to determine the optimal therapies for patients with complex femoropopliteal lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years old
2. Patients with Rutherford classification range from 3 to 6
3. If patients with both lower limbs meeting the inclusion criteria, both side of limb can be selected for this study
4. The lower extremity artery needs to have a healthy runoff of no less than 10 cm above the ankle
5. The guide wire should pass through the lesion of femoropopliteal artery, and further endovascular treatment is performed. In this study, we did not limit the methods of the guide wire passing through the target lesion
6. If the first-time endovascular treatment is failure, patients undergo endovascular treatment successfully at the second time, the patients can still be enrolled
7. For patients with aortoiliac artery lesions, they can be enrolled after the successful reconstruction of aortoiliac artery
8. Informed consent signed by patients

Exclusion Criteria:

1. Patients who are unwilling or refuse to sign the informed consent form
2. Patients with acute and subacute lower extremity arterial thrombosis or arterial embolism
3. Patients with thromboangiitis obliterans
4. Patients with failure of endovascular treatment, and transferred to bypass surgery
5. Patients who underwent surgical atherectomy for common femoral artery occlusive lesions
6. Patients with known allergy to heparin, low molecular weight heparin and contrast agents
7. Patients who have been enrolled in other clinical trials in the past 3 months
8. Women during pregnancy and lactation
9. Patients with other diseases that may lead to difficulties in the trial or significantly shorten the life expectancy (< 3 years), such as tumors, severe liver disease, cardiac insufficiency

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with TASC C, D femoropopliteal lesions who undergoing endovascular treatment
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Technical success rate | 7 days
  Technical success refers to 1. Establishment of continuous blood flow, no early occlusion, acute thrombosis or reintervention driven by target lesion within 7 days after operation
Incidence of major adverse events | 36 months
  major adverse events
Target vessel patency rate evaluated by postoperative ultrasound | 36 months
  Target vessel patency rate
Clinical-driven Target lesion reintervention rate | 36 months
  Target lesion reintervention rate

SECONDARY OUTCOMES:
Clinical-driven Target lesion reintervention rate | 24 months
  Target lesion reintervention rate
Direct medical expenses (3-year cumulative hospitalization expenses and endovascular expenses related to target lesions) | 36 months
  Direct medical expenses

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China